CLINICAL TRIAL: NCT03880266
Title: A Phase 2, Randomized, Double-blind, Vehicle-controlled Efficacy and Safety Study of Glycopyrronium Cloth, 2.4% in Patients With Palmar Hyperhidrosis
Brief Title: A Study of Glycopyrronium Cloth, 2.4% in Patients With Palmar Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM04-HH10
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Palmar Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1 Active (Active Comparator): Glycopyrronium cloth, 2.4% applied to the hands once daily for 14 days: 15 minutes with occlusion (non-latex glove)
  Interventions: Drug: Glycopyrronium cloth, 2.4%
- Group 1 Vehicle (Placebo Comparator): Vehicle cloth applied to the hands once daily for 14 days: 15 minutes with occlusion (non-latex glove)
  Interventions: Drug: Vehicle
- Group 2 Active (Active Comparator): Glycopyrronium cloth, 2.4% applied to the hands once daily for 14 days: 30 minutes with occlusion (non-latex glove)
  Interventions: Drug: Glycopyrronium cloth, 2.4%
- Group 2 Vehicle (Placebo Comparator): Vehicle cloth applied to the hands once daily for 14 days: 30 minutes with occlusion (non-latex glove)
  Interventions: Drug: Vehicle
- Group 3 Active (Active Comparator): Glycopyrronium cloth, 2.4% applied to the hands once daily for 14 days: 15 minutes
  Interventions: Drug: Glycopyrronium cloth, 2.4%
- Group 3 Vehicle (Placebo Comparator): Vehicle cloth applied to the hands once daily for 14 days: 15 minutes
  Interventions: Drug: Vehicle
- Group 4 Active (Active Comparator): Glycopyrronium cloth, 2.4% applied to the hands once daily for 14 days: 30 minutes
  Interventions: Drug: Glycopyrronium cloth, 2.4%
- Group 4 Vehicle (Placebo Comparator): Vehicle cloth applied to the hands once daily for 14 days: 30 minutes
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Glycopyrronium cloth, 2.4% — Pre-saturated 100% polypropylene, nonwoven, fabric cloth with glycopyrronium
  Arms: Group 1 Active; Group 2 Active; Group 3 Active; Group 4 Active
Drug: Vehicle — Pre-saturated 100% polypropylene, nonwoven, fabric cloth
  Arms: Group 1 Vehicle; Group 2 Vehicle; Group 3 Vehicle; Group 4 Vehicle

SUMMARY:
The objective of this study is to assess the efficacy and safety of glycopyrronium cloth, 2.4% when used to treat palmar hyperhidrosis.

DETAILED DESCRIPTION:
This is a pilot study assessing the safety and efficacy of glycopyrronium cloth in patients with palmar hyperhidrosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and assent (for subjects under legal adult age).
2. Age ≥9 years.
3. Primary palmar hyperhidrosis for at least 6 months duration.
4. Average sweat severity score of ≥4 at Baseline.
5. Hyperhidrosis Disease Severity Scale of 3 or 4 at Baseline.
6. Willing to comply with the protocol. Subjects under legal adult age will be assessed by the investigator as to their ability to comply with the protocol.
7. Male or non-pregnant (negative urine pregnancy test in female subjects of child-bearing potential), non-lactating females.

Exclusion Criteria:

1. Subjects who have taken or are currently taking glycopyrronium cloth, 2.4%.
2. Prior surgical procedure for hyperhidrosis.
3. Iontophoresis for the palms within 4 weeks of Baseline.
4. Treatment with botulinum toxin (e.g., Botox®) for palmar hyperhidrosis within 1 year of Baseline.
5. Open wounds or inflammatory lesions on the hands or, any condition that may alter the barrier function of the skin on the hands.
6. Secondary palmar hyperhidrosis or presence of a condition that may cause secondary hyperhidrosis (e.g., lymphoma, malaria, severe anxiety not controlled by medication, carcinoid syndrome, substance abuse, hyperthyroidism).
7. Known history of Sjögren's syndrome or Sicca syndrome.
8. History of glaucoma, inflammatory bowel disease, toxic megacolon, active febrile illness, paralytic ileus, unstable cardiovascular status in acute hemorrhage, severe ulcerative colitis, toxic megacolon complicating ulcerative colitis or myasthenia gravis.
9. Men with a history of urinary retention requiring catheterization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Doherty, Study Director — Dermira, Inc.
Locations (7):
- United States (7):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - International Dermatology Research, Inc., Miami, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Saint Louis University Dermatology, St Louis, Missouri
  - Innovative Dermatology/ ACRC Trials, Plano, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Started | 12 | 6 | 12 | 4 | 12 | 6 | 13 | 7
Completed | 12 | 5 | 11 | 4 | 12 | 6 | 13 | 7
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Vehicle: Vehicle applied to the hands once daily for 14 days: 15 minutes with occlusion (non-latex glove)
- Group 2 Vehicle: Vehicle applied to the hands once daily for 14 days: 30 minutes with occlusion (non-latex glove)
- Group 3 Vehicle: Vehicle applied to the hands once daily for 14 days: 15 minutes
- Group 4 Vehicle: Vehicle applied to the hands once daily for 14 days: 30 minutes
- Total: Total of all reporting groups
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle | Total
Number analyzed (Participants) | 12 | 6 | 12 | 4 | 12 | 6 | 13 | 7 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (8.95) | 34.5 (15.93) | 29.2 (11.57) | 47.5 (17.56) | 28.2 (12.45) | 32.5 (7.97) | 26.6 (9.54) | 37.1 (13.91) | 31.1 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 7 | 4 | 8 | 3 | 8 | 5 | 47
  Male | 4 | 2 | 5 | 0 | 4 | 3 | 5 | 2 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 8
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 8 | 4 | 7 | 4 | 9 | 4 | 12 | 5 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 12 | 4 | 12 | 6 | 13 | 7 | 72
Hand Sweat Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Hand Sweat Severity Score is a patient reported outcome, designed to measure the severity of palmar hyperhidrosis [score on a scale from 0 (better) -10 (worse)].
  units on a scale | 6.78 (1.646) | 7.40 (0.718) | 7.56 (1.450) | 8.10 (1.920) | 6.93 (1.689) | 7.37 (2.017) | 7.58 (1.399) | 8.01 (1.078) | 7.37 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 2 in Hand Sweating Severity Score
Description: The Hand Sweat Severity Score is a patient reported outcome, designed to measure the severity of palmar hyperhidrosis [score on a scale from 0 (better) -10 (worse)].
Time Frame: Baseline, Week 2
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Number analyzed (Participants) | 12 | 5 | 11 | 4 | 12 | 6 | 13 | 7
score on a scale | -2.14 (2.199) | -0.56 (0.730) | -1.64 (1.410) | -3.03 (2.161) | -2.53 (2.223) | -2.20 (1.084) | -1.30 (2.062) | -1.34 (1.909)
Statistical Analysis 1: Comparison: Group 1 Active vs Group 1 Vehicle; Test type: Superiority; p = 0.244, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-3.76 to 0.60]
Statistical Analysis 2: Comparison: Group 2 Active vs Group 2 Vehicle; Test type: Superiority; p = 0.168, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-0.65 to 3.43]
Statistical Analysis 3: Comparison: Group 3 Active vs Group 3 Vehicle; Test type: Superiority; p = 0.699, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-2.39 to 1.72]
Statistical Analysis 4: Comparison: Group 4 Active vs Group 4 Vehicle; Test type: Superiority; p = 0.833, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.94 to 2.02]

2. Secondary Outcome: Percentage of Subjects Who Have a ≥2 Grade Improvement in HDSS (Hyperhidrosis Disease Severity Scale) From Baseline at Week 2
Description: Hyperhidrosis Disease Severity Scale (HDSS) is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.
  1 (better), 2, 3, 4 (worse)
Time Frame: Baseline, Week 2
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Number analyzed (Participants) | 12 | 5 | 10 | 4 | 11 | 6 | 13 | 7
Participants | 3 | 0 | 1 | 2 | 1 | 2 | 3 | 2
Statistical Analysis 1: Comparison: Group 1 Active vs Group 1 Vehicle; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Group 2 Active vs Group 2 Vehicle; Test type: Superiority; p = 0.589, Fisher Exact
Statistical Analysis 3: Comparison: Group 3 Active vs Group 3 Vehicle; Test type: Superiority; p = 0.154, Fisher Exact
Statistical Analysis 4: Comparison: Group 4 Active vs Group 4 Vehicle; Test type: Superiority; p = 0.646, Fisher Exact

3. Secondary Outcome: Mean Absolute Change From Baseline in Gravimetrically-measured Sweat Production at Week 2
Description: Gravimetrically measured sweat production is based on the mean of the right and left hand measurements; average of the change in the gravimetric measurement of sweat produced at baseline compared with Week 2
Time Frame: Baseline, Week 2
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Number analyzed (Participants) | 12 | 5 | 11 | 4 | 12 | 6 | 13 | 7
mg | -69.8 (162.54) | 136.7 (320.57) | -15.3 (53.14) | -159.4 (354.38) | -113.5 (164.10) | 38.1 (106.30) | -58.6 (139.70) | 102.0 (767.52)
Statistical Analysis 1: Comparison: Group 1 Active vs Group 1 Vehicle; Test type: Superiority; p = 0.093, t-test, 2 sided; Mean Difference (Final Values) = -206.5, 95% CI 2-sided [-451.9 to 38.9]
Statistical Analysis 2: Comparison: Group 2 Active vs Group 2 Vehicle; Test type: Superiority; p = 0.186, t-test, 2 sided; Mean Difference (Final Values) = 144.1, 95% CI 2-sided [-78.6 to 366.7]
Statistical Analysis 3: Comparison: Group 3 Active vs Group 3 Vehicle; Test type: Superiority; p = 0.058, t-test, 2 sided; Mean Difference (Final Values) = -151.7, 95% CI 2-sided [-309.0 to 5.7]
Statistical Analysis 4: Comparison: Group 4 Active vs Group 4 Vehicle; Test type: Superiority; p = 0.186, t-test, 2 sided; Mean Difference (Final Values) = 160.6, 95% CI 2-sided [-611.2 to 290.1]

4. Secondary Outcome: Mean Percent Change From Baseline in Gravimetrically-measured Sweat Production at Week 2
Description: Gravimetrically measured sweat production is based on the mean of the right and left hand measurements; calculation of percentage difference in sweat production at week 2 compared to baseline sweat production
Time Frame: Baseline, Week 2
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Number analyzed (Participants) | 12 | 5 | 11 | 4 | 12 | 6 | 13 | 7
Percent change | -17.1 (28.26) | 16.5 (60.4) | -7.5 (65.53) | -31.8 (51.29) | -26.8 (39.17) | 11.4 (34.96) | -17.7 (40.43) | 21.7 (145.81)
Statistical Analysis 1: Comparison: Group 1 Active vs Group 1 Vehicle; Test type: Superiority; p = 0.130, t-test, 2 sided; Mean Difference (Final Values) = -33.62, 95% CI 2-sided [-78.42 to 11.17]
Statistical Analysis 2: Comparison: Group 2 Active vs Group 2 Vehicle; Test type: Superiority; p = 0.518, t-test, 2 sided; Mean Difference (Final Values) = 24.26, 95% CI 2-sided [-54.62 to 103.13]
Statistical Analysis 3: Comparison: Group 3 Active vs Group 3 Vehicle; Test type: Superiority; p = 0.061, t-test, 2 sided; Mean Difference (Final Values) = -38.14, 95% CI 2-sided [-78.32 to 2.03]
Statistical Analysis 4: Comparison: Group 4 Active vs Group 4 Vehicle; Test type: Superiority; p = 0.366, t-test, 2 sided; Mean Difference (Final Values) = -39.34, 95% CI 2-sided [-128.40 to 49.72]

5. Secondary Outcome: Percentage of Subjects Who Have at Least a 50% Reduction in Gravimetrically-measured Sweat Production From Baseline at Week 2
Description: Gravimetrically measured sweat production is based on the mean of the right and left hand measurements; confidence interval represents difference between vehicle and active group
Time Frame: Baseline, Week 2
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
Number analyzed (Participants) | 12 | 5 | 11 | 4 | 12 | 6 | 13 | 7
Participants | 1 | 1 | 3 | 2 | 4 | 0 | 2 | 3
Statistical Analysis 1: Comparison: Group 1 Active vs Group 1 Vehicle; Test type: Superiority; p = 0.515, Fisher Exact
Statistical Analysis 2: Comparison: Group 2 Active vs Group 2 Vehicle; Test type: Superiority; p = 0.560, Fisher Exact
Statistical Analysis 3: Comparison: Group 3 Active vs Group 3 Vehicle; Test type: Superiority; p = 0.245, Fisher Exact
Statistical Analysis 4: Comparison: Group 4 Active vs Group 4 Vehicle; Test type: Superiority; p = 0.290, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through Week 2
Description: All subjects who are randomized and receive at least one confirmed dose of study drug will be included in the safety population.
Arm/Group | Group 1 Active | Group 1 Vehicle | Group 2 Active | Group 2 Vehicle | Group 3 Active | Group 3 Vehicle | Group 4 Active | Group 4 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/12 | 0/4 | 0/12 | 0/6 | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/12 | 0/4 | 0/12 | 0/6 | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 5/12 | 2/6 | 5/12 | 1/4 | 1/12 | 2/6 | 2/13 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Active (N=12) | Group 1 Vehicle (N=6) | Group 2 Active (N=12) | Group 2 Vehicle (N=4) | Group 3 Active (N=12) | Group 3 Vehicle (N=6) | Group 4 Active (N=13) | Group 4 Vehicle (N=7)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compensatory sweating (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03880266/Prot_SAP_000.pdf